CLINICAL TRIAL: NCT05277064
Title: Optimal Preliminary Insertion Depth of Fiberoptic Bronchoscope for Visualization of Glottic Opening in Oral Fiberoptic Intubation
Brief Title: Optimal Insertion Depth of FOB for Oral FOB Intubation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jung-Man Lee, Clinical Associate professor, Seoul National University Hospital
Other Study IDs: 10-2021-95
Record Dates: First submitted 2022-01-26; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: General Anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Oral FOB — After induction of anesthesia and muscle relaxation, An investigator who has experiences of numerous fiberoptic intubations will measure the optimal preliminary insertion depth of the fiberoptic bronchoscope for oral fiberoptic intubation.

SUMMARY:
For oral fiberoptic intubation, the preliminary insertion depth of the fiberoptic bronchoscope should be important because the excessive insertion depth or too shallow depth might be the reason why the clinicians cannot perform oral fiberoptic intubation completely.

The purpose of the study is to find out the optimal preliminary insertion depth of the fiberoptic bronchoscope for visualization of glottic opening in oral fiberoptic intubation.

DETAILED DESCRIPTION:
For oral fiberoptic intubation, the preliminary insertion depth of the fiberoptic bronchoscope should be important because the excessive insertion depth or too shallow depth might be the reason why the clinicians cannot perform oral fiberoptic intubation completely.

The purpose of the study is to find out the optimal preliminary insertion depth of the fiberoptic bronchoscope for visualization of glottic opening in oral fiberoptic intubation.

The investigators will enroll the subjects of the present study after obtaining the written consent.

After enrollment, the investigators will measure some anatomical distance, such as patient height.

After induction of anesthesia and muscle relaxation for tracheal intubation, An investigator who has experiences of numerous fiberoptic intubation will measure the optimal preliminary insertion depth of the fiberoptic bronchoscope from the philtrum, the upper lip, or the incisors for oral fiberoptic intubation, with the aid of assistants. Then, tracheal intubation with a laryngoscope as a routine manner of our institute.

The investigators will calculate the mean value of the optimal depth and find out an formula for that from our data.

ELIGIBILITY:
Inclusion Criteria:

* patients requiring tracheal intubation for general anesthesia

Exclusion Criteria:

* do not agree to participate in the study
* emergency surgery
* predicted difficult intubation
* very weak teeth (especially central teeth)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients requiring tracheal intubation for general anesthesia without exclusion criteria of our study
Sampling Method: Non-Probability Sample
Enrollment: 211 (Estimated)
Dates: Start 2022-03-07 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
The length of optimal preliminary insertion depth of FOB (centimeters) | during tracheal intubation
  The length of optimal preliminary insertion depth of FOB means the insertion depth of it from the philtrum, the upper lip, or the incisors where the clinicians can see easily the glottic opening while they are flexing the FOB. And that will be recorded as centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Man Lee, MD.PhD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
If there will be a reasonable request, we will provide the study data after approval of that from the IRB of our institute.